CLINICAL TRIAL: NCT01271244
Title: Effects of Escitalopram on Autonomic Reactivity in Post Traumatic Stress Disorder Among Veterans of Operation Enduring Freedom and Iraqi Freedom (OEF/OIF)
Brief Title: Effects of Escitalopram on Autonomic Reactivity in Post Traumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Sriram Ramaswamy, Staff Psychiatrist, VA Nebraska Western Iowa Health Care System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAM 6-7-2008
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTSD Depression Group (Active Comparator): Escitalopram 10-20 mg/day
  Interventions: Drug: Escitalopram
- Major Depression Group (Active Comparator): Escitalopram 10-20 mg/day
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10-20mg daily for 12 weeks
  Other Names: Lexapro

SUMMARY:
The study looked at relationship between escitalopram and heart rate variability and QT variability in veterans with PTSD.

DETAILED DESCRIPTION:
The investigators are studying if taking escitalopram will normalize heart rate variability and a decrease (or no effect implying a lack of serious cardiac side effects) including QT variability in veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - Group I
* Patients, men and women between 19 and 55 years of age, inclusive.
* Patients with diagnosis of Posttraumatic Stress Disorder as determined by Mini-International Neuropsychiatric Interview (M.I.N.I.).
* Patients, who are able to comprehend and satisfactorily comply with protocol requirements and have an ability to read and write English.
* Patients, who signed the written informed consent given prior to entering any study procedure.
* Inclusion Criteria - Group II
* Patients, men and women between 19 and 55 years of age, inclusive.
* Patients with diagnosis of Major Depression as determined by Mini-International Neuropsychiatric Interview (M.I.N.I.). A diagnosis of PTSD will be exclusionary.
* Patients, who are able to comprehend and satisfactorily comply with protocol requirements and have an ability to read and write English.
* Patients, who signed the written informed consent given prior to entering any study procedure.

Exclusion Criteria:

* History of cardiovascular disease or a history of hypertension.
* Patients with a concurrent Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis in any of the following categories as determined by the M.I.N.I.
* Lifetime Schizophrenia and Schizoaffective Disorder
* Lifetime Bipolar I Disorder
* Substance Dependence or Abuse (excluding nicotine) within one month prior to the Screening Visit.
* Patients with a history of intolerance or hypersensitivity to escitalopram or citalopram.
* Patients who based on history or mental status examination have a significant risk of committing suicide. Current suicide risk (past month) will be assessed using the M.I.N.I. Suicidality Module. Subjects considered at high suicide risk based on the module (> 17 points) will be excluded from study participation.
* Patients who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
* Subjects will be excluded who have a history of significant medical illness and who are on medications that affect cardiac and/or autonomic function.
* Female patients who are pregnant, planning to become pregnant, or if of childbearing potential, not using an acceptable method of birth control.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, MD, Principal Investigator — Department of Veterans Affairs/NWIHCS
Locations (1):
- Omaha Veterans Affairs Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PTSD Depression Group: Veterans with PTSD and depression will receive Escitalopram: 10-20mg daily for 12 weeks
- Major Depression Group: Veteran with Depression only will receive Escitalopram: 10-20mg daily for 12 weeks
Period: Overall Study
Arm/Group | PTSD Depression Group | Major Depression Group
Started | 18 | 8
Completed | 11 | 5
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Major Depression Group: Veterans with Depression only will receive Escitalopram: 10-20mg daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | PTSD Depression Group | Major Depression Group | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 28.3 (2.4) | 30 (4.1) | 29 (1.41)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 11 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: High Frequency Heart Rate Variability
Description: Heart rate variability is the standard deviation of successive R-to-R intervals, or variability in time between successive heart beats. Spectral power in the high frequency (HF: 0.15-0.5 Hz) band reflects parasympathetic input, or cardiac vagal function. A natural log (ln) transformation was applied to heart rate variability data to derive the outcome measure.
Time Frame: 12 Weeks
Population: Due to the small number of subjects in the major depression group, results were not analyzed for this group.
Measure: Mean (Standard Deviation); unit: ln(msec)
Groups:
- PTSD Depression Group: Veterans with PTSD and depression receive Escitalopram: 10-20mg daily for 12 weeks
- Major Depression Group: Veterans with major depression receive Escitalopram: 10-20mg daily for 12 weeks
Arm/Group | PTSD Depression Group | Major Depression Group
Number analyzed (Participants) | 11 | 0
ln(msec)
  Pre-treatment | 6.31 (1.16) |
  Post-treatment | 5.48 (0.67) |

2. Primary Outcome: QT Interval Variability
Description: QT variability index (QTvi) is a measure of QT variability normalized to heart rate variability. Increased QTvi has been associated with increased sympathetic activity. QTvi was calculated using Berger's formula as the log ratio of QT variability normalized by the squared mean QT interval divided by heart rate variability normalized by the squared mean heart rate. QTvi is normally expressed as a negative value, and a less negative QTvi may reflect increased QT variability or reduced heart rate variability.
Time Frame: 12 weeks
Population: Due to the small number of subjects in the major depression group, results were not analyzed for this group.
Measure: Mean (Standard Deviation); unit: log ratio
Arm/Group | PTSD Depression Group | Major Depression Group
Number analyzed (Participants) | 11 | 0
log ratio
  Pre-treatment | -1.82 (0.43) |
  Post-treatment | -1.32 (0.67) |

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Major Depression Group: Veterans with Major Depression only receive Escitalopram: 10-20mg daily for 12 weeks
Arm/Group | PTSD Depression Group | Major Depression Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/8
Other Adverse Events (participants affected / at risk) | 0/18 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTSD Depression Group (N=18) | Major Depression Group (N=8)
Suicidal Ideation (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to small number of subjects recruited in major depression group we are unable to compare to the PTSD group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No